CLINICAL TRIAL: NCT02501590
Title: Differences in Muscle Activity Patterns and Graphical Product Quality in Children With Graphomotor Impairment Copying and Tracing Activities on Horizontal or Vertical Surfaces
Brief Title: Differences in Muscle Activity Patterns and Graphical Product Quality in Children With Graphomotor Impairment
Status: Completed | Type: Observational
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, Aviva Mimouni-Bloch, Head of The Pediatric Neurology and Developmental Unit, Loewenstein Hospital
Other Study IDs: 22-14-LOE
Record Dates: First submitted 2015-07-08; First posted 2015-07-17 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Graphomotor Impairment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- study: After the parents sign an informed consent form, they will fill out a demographic questionnaire. Than if the Beery VMI test was not yet administered, it would be performed, as well as the Developmental Coordination Disorder Questionnaire (DCD-Q). Surface electromyography electrodes will be placed on the Upper Trapezius, Extensor Carpi Radialis, and Biceps brachii of the child's dominant hand.
  The subject will perform 4 copying tasks and 2 tracing tasks on a tablet placed once on a horizontal surface (while sitting) and once on a vertical surface (while standing).
- control: After the parents sign an informed consent form, they will fill out a demographic questionnaire. Than if the Beery VMI test was not yet administered, it would be performed, as well as the Developmental Coordination Disorder Questionnaire (DCD-Q). Surface electromyography electrodes will be placed on the Upper Trapezius, Extensor Carpi Radialis, and Biceps brachii of the child's dominant hand.
  The subject will perform 4 copying tasks and 2 tracing tasks on a tablet placed once on a horizontal surface (while sitting) and once on a vertical surface (while standing).

SUMMARY:
Drawing on a vertical surface, rather than horizontal (such as blackboard) is often used by occupational therapists as a way of developing fine motor control and visual motor integration in children. In healthy children no difference in graphical quality was shown between drawing on vertical or horizontal surfaces. However, this was not investigated in children with graphomotor impairments.

The goal of this study is to determine whether movements produced on a vertical surface differ in their performance level and muscle activation patterns compared to movements produced on a horizontal surface. The investigators predict that there would be a difference in the level of performance between the two surfaces.

DETAILED DESCRIPTION:
Drawing on a vertical surface, such as a blackboard (rather than a horizontal surface) is often used by occupational therapists as a way of developing fine motor control and visual motor integration in children. While there is anecdotal evidence to support this intervention, preliminary results in healthy children showed no differences in graphical quality while drawing on vertical or horizontal surfaces. This however was not investigated in children with graphomotor impairments.

The goal of this study is to determine whether movements produced on a vertical surface differ in their performance level and muscle activation patterns compared to movements produced on a horizontal surface.

The investigators predict that the level of performance on the vertical surface will exceed the level of performance on the horizontal surface. Additionally, the investigators hypothesize that the proximal muscles will be more activated and fatigued (in longer tasks) while drawing on the vertical surface, while the distal muscle will be more activated and fatigued while drawing on the horizontal surface.

ELIGIBILITY:
Study group Inclusion criteria:

* Up to 50 percentile in the long form Beery-Buktenica Developmental Test of Visual-Motor Integration (Beery VMI).

Exclusion Criteria:

* children in special education,
* any orthopedic or neurologic impairment,
* visual impairment that could not be corrected with glasses, or
* ability to understand and follow simple instructions, reported by the parents.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of Forty five 4-6 years old children, referred to occupational therapy
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aviva Mimouni-Bloch, M.D, Principal Investigator — Clalit Health Services
Locations (2):
- Israel (2):
  - Loewenstein hospital, Raanana
  - Loewenstein Rehabilitation Center, Raanana

REFERENCES:
- [Background] McHale K, Cermak SA. Fine motor activities in elementary school: preliminary findings and provisional implications for children with fine motor problems. Am J Occup Ther. 1992 Oct;46(10):898-903. doi: 10.5014/ajot.46.10.898. PMID 1463061
- [Background] Schwellnus H, Carnahan H, Kushki A, Polatajko H, Missiuna C, Chau T. Effect of pencil grasp on the speed and legibility of handwriting after a 10-minute copy task in Grade 4 children. Aust Occup Ther J. 2012 Jun;59(3):180-7. doi: 10.1111/j.1440-1630.2012.01014.x. PMID 22690768
- [Background] Ratzon NZ, Efraim D, Bart O. A short-term graphomotor program for improving writing readiness skills of first-grade students. Am J Occup Ther. 2007 Jul-Aug;61(4):399-405. doi: 10.5014/ajot.61.4.399. PMID 17685172
- [Background] Yakimishyn JE, Magill-Evans J. Comparisons among tools, surface orientation, and pencil grasp for children 23 months of age. Am J Occup Ther. 2002 Sep-Oct;56(5):564-72. doi: 10.5014/ajot.56.5.564. PMID 12269511
- [Background] Wilson BN, Kaplan BJ, Crawford SG, Campbell A, Dewey D. Reliability and validity of a parent questionnaire on childhood motor skills. Am J Occup Ther. 2000 Sep-Oct;54(5):484-93. doi: 10.5014/ajot.54.5.484. PMID 11006808

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study | Control
Started | 13 | 35
Completed | 13 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study | Control | Total
Number analyzed (Participants) | 13 | 35 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 35 | 48
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.9 (0.5) | 5.9 (0.4) | 5.4 (0.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 18 | 22
  Male | 9 | 17 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 13 | 35 | 48

OUTCOME MEASURES:

1. Primary Outcome: Normilized Muscle Activity
Description: The maximal voluntary contraction (MVC) value for each muscle will be computed as the average of three peaks of the surface electromyography (sEMG) data, which differed by no more than 10% from one another. The mean root mean square (RMS) values of the sEMG data will be normalized by the MVC value for each muscle so that the value is presented by percentage.
Time Frame: day1
Measure: Median (Inter-Quartile Range); unit: % mvc
Arm/Group | Study | Control
Number analyzed (Participants) | 13 | 35
% mvc | 8.20 [4.75 to 18.78] | 7.41 [5.58 to 9.69]
Statistical Analysis 1: Comparison: Study vs Control; Test type: Other; p = 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Study | Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/35
Other Adverse Events (participants affected / at risk) | 0/13 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No